CLINICAL TRIAL: NCT00744224
Title: Prednisolone-induced Impairment of Glucose Metabolism and Beta-cell Dysfunction and the Protective Effects of Exenatide: a Single-center, Randomized, Double-blind, Placebo-controlled Crossover Study in Healthy Volunteers
Brief Title: PREDnisolone-induced Beta-cell Dysfunction Prevented by EXenatide
Acronym: PREDEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: National Research Council, Institute of Biomedical Engineering (Unknown)
Responsible Party: Dr M Diamant, VU University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DC2008pred003
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Glucocorticoid-induced Glucometabolic Abnormalities; Glucocorticoid-induced Beta-cell Dysfunction
MeSH Terms: interventions — Prednisolone; Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Prednisolone
- 3 (Active Comparator)
  Interventions: Drug: Prednisolone and Exenatide

INTERVENTIONS:
Drug: Placebo — Single dose of placebo with saline infusion
  Arms: 1
Drug: Prednisolone — Single dose of 80 mg prednisolone with saline infusion
  Arms: 2
Drug: Prednisolone and Exenatide — Prednisolone 80 mg single dose Exenatide infusion 20 mg/min
  Arms: 3

SUMMARY:
The purpose of this study is to explore whether the GLP-1 receptor agonist exenatide, may prevent glucocorticoid-induced glucometabolic abnormalities and beta-cell dysfunction in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* 18 years ≤ age ≤ 35 years on the day of the first visit
* 22.0 ≤ BMI ≤ 28.0 kg/m2
* (History of) good physical and mental health as determined by history taking, physical and laboratory examinations and ECG.
* fasting glucose level of < 5.6 mmol/L, in addition to a glucose level of < 7.8 mmol/L at 2 hours after intake of 75 g glucose (OGTT).
* able to keep a normal day and night rhythm during the trial period (i.e. no shift work)

Exclusion Criteria:

* history or presence of a medical disorder
* use of drugs, except for incidental (non-opioid) analgesic agents
* first degree relative with T2DM
* performing intensive physical activity > 1x/week
* an allergic or anaphylactic reaction to prednisolone treatment in the past
* clinically relevant history or presence of any medical disorder, which are mentioned in the Summary of Product Characteristics (SPC) as contraindication for the use of prednisolone
* glucocorticosteroid use during the last three months prior to the first dose
* participation in an investigational drug trial within 90 days prior to the first dose
* donation of blood (> 100 mL) within 90 days prior to the first dose
* history of or current abuse of drugs or alcohol (>14 U/week)
* smoking
* use of grapefruit products during the study period
* recent changes in weight and/or physical activity
* serious mental impairment or language problems i.e. preventing to understand the study protocol/aim

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To assess whether a single day infusion of the GLP-1 RA exenatide, as compared to placebo, reverses GC-induced impairment of glucose metabolism in healthy males, quantified as glucose tolerance (AUCgluc) during a standardized mixed-meal test | Single-day treatment

SECONDARY OUTCOMES:
To assess whether a single day infusion of the GLP-1 RA exenatide, as compared to placebo, reverses GC-induced acute beta-cell dysfunction in healthy males, quantified as Various measures of beta-cell function | Single day treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Diamant, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van Raalte DH, van Genugten RE, Linssen MM, Ouwens DM, Diamant M. Glucagon-like peptide-1 receptor agonist treatment prevents glucocorticoid-induced glucose intolerance and islet-cell dysfunction in humans. Diabetes Care. 2011 Feb;34(2):412-7. doi: 10.2337/dc10-1677. Epub 2011 Jan 7. PMID 21216851